CLINICAL TRIAL: NCT02669173
Title: Targeting Myeloid Derived Suppressor Cells in Recurrent Glioblastoma: Phase 0/1 Trial of Low Dose Capecitabine + Bevacizumab in Patients With Recurrent Glioblastoma
Brief Title: Capecitabine + Bevacizumab in Patients With Recurrent Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE7315
Record Dates: First submitted 2016-01-21; First posted 2016-02-01 (Estimated); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Glioblastoma
Keywords: Myeloid derived suppressor cells; brain tumor; MDSC; GBM; recurrent
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Recurrence | interventions — Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment: Capecitabine + Bevacizumab (Experimental): Capecitabine, PO dose to be determined by phase 1 dose escalation, cycle length 28 days. Treated with Bevacizumab, IV, 10 mg/kg days 1, 15 every 28 days, until progression.
  Interventions: Drug: Capecitabine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Capecitabine — Drug given orally. Dose to be determined by phase 1 dose escalation, cycle length 28 days. Treatment until progression
Drug: Bevacizumab — Drug given by IV, 10 mg/kg days 1, 15 every 28 days, until progression.

SUMMARY:
This study involves participants with recurrent glioblastoma brain tumors (GBM). This means that a participant's brain tumor has either returned after being treated by a previous therapy, or has continued to progress despite being treated.

The purpose of this study is to provide proof of concept that suppression of MDSCs (myeloid-derived suppressor cells) is feasible in patients with GBM. Rather than targeting tumor cells or immune checkpoints, which has been the focus of recent therapeutic efforts, direct targeting of MDSCs with low dose capecitabine has the potential to reverse the immunosuppressed microenvironment of GBM and thereby reduce tumors

DETAILED DESCRIPTION:
Primary Objective: To achieve a 20-fold MDSC reduction in the concentration of circulating MDSCs after treatment with low dose capecitabine.

Secondary Objectives:

1. To determine the concentration of circulating MDSCs in patients with recurrent glioblastoma after treatment with low dose capecitabine
2. To determine the concentration of tissue MDSCs and T-regulatory cells in resected glioblastoma after treatment with low dose capecitabine
3. To determine the safety and toxicity of continuous low dose capecitabine with and without standard dose bevacizumab.

Exploratory Objective:

To obtain a signal for efficacy as measured by progression-free survival rate at 6 months

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed WHO grade 4 glioma for which a clinically indicated tumor resection is planned.
* Subjects must not have received capecitabine or bevacizumab for this disease.
* Performance status: Karnofsky Performance status ≥ 60%
* Subjects must have adequate organ function and laboratory parameters within 21 days of study entry as defined below:

  * Hemoglobin ≥ 8 g/dl
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelet count ≥ 100,000/mcL
  * Total bilirubin < 1.5 x institutional upper limit of normal (ULN)
  * AST (SGOT) ≤ 3 X institutional ULN
  * ALT (SGPT) ≤ 3 X institutional ULN
  * Calculated creatinine clearance ≥ 50 mL/min
  * Urine protein screened by urine analysis for urine protein creatinine (UPC) ratio. For UPC ratio > 0.5, 24-hour urine protein must be obtained and must be < 1000 mg.
  * Prothrombin time/international normalized ratio (PT/INR) < 1.4 for patients not on warfarin
  * Patients on full-dose anticoagulants (e.g., warfarin or LMW heparin) must meet both of the following criteria:

    * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
    * In-range international normalized ratio (between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* Women of childbearing potential must have a negative pregnancy test within 21 days of study entry. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and through 30 days after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and through 30 days after the last dose of study drug.
* Patients must be able to swallow whole tablets.
* Systolic blood pressure ≤ 160 mg Hg or diastolic pressure ≤ 90 mg Hg within 14 days prior to study registration
* Electrocardiogram without evidence of acute cardiac ischemia within 14 days prior study registration
* Patients must have the following minimum intervals from prior treatments:

  * surgery - 4 weeks
  * nitrosoureas - 6 weeks
  * cytotoxic chemotherapy - standard intervals depending on the most recent regimen. i.e., for temozolomide 5 of 28, 23 days after most recent temozolomide; for temozolomide 21 of 28 days, 7 days after most recent dose; etoposide 14 of 21 days, 7 days after last dose. For drugs not listed, the research nurse, treating investigator, and principal investigator will determine the appropriate interval.
  * Investigational therapy or non cytotoxic therapy - 2 weeks

Exclusion Criteria:

* Prior treatment toxicities not resolved to ≤ Grade 1 according to NCI CTCAE Version 4.0 except alopecia and neuropathy.
* Subjects receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to capecitabine or bevacizumab.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive subjects on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with capecitabine and/or bevacizumab. In addition, these subjects are at increased risk of lethal infections when treated with marrow suppressive therapy.
* Other malignancy within the past 2 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or vulva; c) prostate cancer of Gleason Score 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder, or benign tumors of the adrenal or pancreas.
* Significant chronic gastrointestinal disorder with diarrhea as a major symptom (e.g., Crohn's disease, malabsorption, or Grade ≥2 (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events Version 4.0 [CTCAE v.4.0] diarrhea of any etiology at screening).
* Active infection with hepatitis B or hepatitis C virus.
* Pregnant or breastfeeding.
* Known dihydropyrimidine dehydrogenase deficiency.
* Known hypersensitivity to 5-fluorouracil, capecitabine, bevacizumab or to any component of the investigational products or compounds of similar chemical composition.
* Unable or unwilling to swallow tablets.
* Evidence of significant medical illness, abnormal laboratory finding, or psychiatric illness/social situations that would, in the Investigator's judgment, make the patient inappropriate for this study.
* Arterial ischemic event (e.g., unstable angina, myocardial infarction, stroke) within 6 months of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change of concentration in circulating MDSCs after treatment with low dose capecitabine | baseline to eight months after

SECONDARY OUTCOMES:
Concentration of MDSCs in resected glioblastoma after treatment with low dose capecitabine | Eight months
Concentration of T-regulatory cells after treatment with low dose capecitabine | Eight months
Number of participants with adverse events relating to treatment with low-dose capecitabine alone as assessed by CTCAE v4.0 | Nine months
Number of participants with adverse events relating to treatment with low-dose capecitabine combined with bevacizumab as assessed by CTCAE v4.0 | Nine months

OTHER OUTCOMES:
To obtain a signal for efficacy as measured by progression-free survival rate at 6 months | Six months

CONTACTS AND LOCATIONS:
Overall Officials: David Peereboom, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Peereboom DM, Alban TJ, Grabowski MM, Alvarado AG, Otvos B, Bayik D, Roversi G, McGraw M, Huang P, Mohammadi AM, Kornblum HI, Radivoyevitch T, Ahluwalia MS, Vogelbaum MA, Lathia JD. Metronomic capecitabine as an immune modulator in glioblastoma patients reduces myeloid-derived suppressor cells. JCI Insight. 2019 Nov 14;4(22):e130748. doi: 10.1172/jci.insight.130748. PMID 31600167